CLINICAL TRIAL: NCT03530449
Title: Evaluation of the Repeatability and Reproducibility of OCTA Image Quality With the Heidelberg Engineering SPECTRALIS With OCT Angiography Module
Status: Terminated | Type: Observational
Why Stopped: Management decision; not patient safety related
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2018-1
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Retinal Vascular; Normal Eyes
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects with Normal Eyes: Color Fundus Photography, Optical Coherence Tomography, and OCT Angiography scans as per protocol in subjects without ophthalmic pathology
  Interventions: Device: OCT Angiography; Device: Color Fundus Photography; Device: Optical Coherence Tomography
- Subjects with Retinal Vascular Pathology: Color Fundus Photography, Optical Coherence Tomography, and OCT Angiography scans as per protocol in subjects with retinal vascular ophthalmic pathology
  Interventions: Device: OCT Angiography; Device: Color Fundus Photography; Device: Optical Coherence Tomography

INTERVENTIONS:
Device: OCT Angiography — OCT Angiography offers clinicians a non-invasive three-dimensional visualization of vasculature in the retina and choroid. The visualization of perfused vasculature in a three-dimensional layout, offers clinicians an aid in the identification of retinal and choroidal pathologies such as retinal ischemia, microaneurysms, retinal neovascularization and choroidal neovascular membranes.
  Other Names: OCTA
Device: Color Fundus Photography — Non-contact white light photography
  Other Names: CFP
Device: Optical Coherence Tomography — Two and Three dimensional cross sectional imaging of the back of the eye to look at vascular structures and is an aid in the detection and management of various ocular diseases.
  Other Names: Structural OCT; OCT

SUMMARY:
Repeatability and Reproducibility of OCTA Image Quality with the Heidelberg Engineering SPECTRALIS

DETAILED DESCRIPTION:
The objectives of this study are to:

1. Assess the repeatability and reproducibility of the SPECTRALIS with OCTA Module image quality
2. Assess the repeatability and reproducibility of visibility of key anatomical vascular structures in the SPECTRALIS with OCTA Module

ELIGIBILITY:
Inclusion Criteria:

* All subjects: Able and willing to undergo the test procedures, sign informed consent, and follow instructions.
* Age ≥ 22

Subjects with Normal Eyes:

* Corrected visual acuity ≥ 20/40 in each eye

Subjects with Pathology:

* Subjects with vascular retinal conditions in at least one eye
* Subjects included should have a range of retinal vascular pathologies likely to appear in OCTA imaging, affecting different anatomic depths through the retina and choroid. Retinal conditions including but not limited to diabetic retinopathy, wet age-related macular degeneration (AMD), and branch or central retinal vein occlusion that give rise to features such as retinal ischemia, microaneurysms, choroidal neovascularization and retinal neovascularization will be included.

Exclusion Criteria:

* All Subjects:
* Subjects unable to read or write
* Subjects with ocular media not sufficiently clear to obtain acceptable study- related imaging
* Subjects who cannot tolerate the imaging procedures
* Subjects with contraindication to pupillary dilation in the study eye
* Subjects with Normal Eyes:
* Subjects with uncontrolled systemic conditions, or ocular disease, as determined by the Investigator, during the eye exam and CFP
* History of ocular surgical intervention (except for refractive or cataract surgery) in either eye

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pathology Population:
  Subjects included should have a range of retinal vascular pathologies likely to appear in OCTA imaging, affecting different anatomic depths through the retina and choroid. Retinal vascular conditions including but not limited to diabetic retinopathy, wet age-related macular degeneration (AMD), and branch or central retinal vein occlusion that give rise to features such as retinal ischemia, microaneurysms, choroidal neovascularization and retinal neovascularization will be included.
  Normal Population:
  In order to be included in the Normal population, subjects will have to meet all inclusion/exclusion criteria for both eyes. Subjects with a history of ocular surgical interventions will be excluded except for those with refractive and/or cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
OCTA image quality | day 1
  Image quality grading results of study selected images
Visualization of key anatomical vascular structures on OCTA | day 1
  Grading of visibility of key anatomical vascular structures of study selected images

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell W Dul, OD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- State University of New York College of Optometry (SUNY), New York, New York, United States